CLINICAL TRIAL: NCT06738134
Title: Implementation of Differentiated Service Delivery Model of Care for People Living with HIV with Comorbidities
Brief Title: Differentiated Service Delivery (DSD) for People Living with HIV (PLHIV) and Comorbidities
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Grace Lui, Clinical Associate Professor (Honorary), Chinese University of Hong Kong
Other Study IDs: DSD_v1_dated 13Mar2024
Record Dates: First submitted 2024-03-20; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Delivery of Health Care; HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is an implementation study evaluating differentiated service delivery model for the care of comorbidities for people living with HIV (PLWH). The Hybrid Type 3 study design is adopted, with the primary goal of evaluating implementation outcomes, and secondary goals of evaluating service and client outcomes according to the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) framework, including Proctor's Conceptual Framework for Implementation Outcomes, using mixed methods for data collection and analyses. PLWH will be identified from the Integrated Treatment Centre, an HIV clinic in Hong Kong, which provides care to around 3500 PLWH, with services including out-patient care of patients with human immunodeficiency virus (HIV) infection, antiviral therapy for HIV and hepatitis co-infection, and treatment of sexually transmitted diseases. PLWH with comorbidities will be asked to participate in a survey for willingness to participate. Those interested will be co-managed at the HIV Comorbidities Clinic at the Prince of Wales Hospital, where the DSD model of care is conducted. Evaluation of implementation outcomes will be performed at the end of the programme.

DETAILED DESCRIPTION:
PLWH who are receiving effective and durable anti-retroviral therapy (ART) have similar life expectancy as the general population, but the patients do suffer from two-fold higher burden of disability associated with chronic comorbidities as compared with people without HIV infection. The screening and management of these chronic comorbidities are gaining attention in both high-income and low- and middle-income settings.

There are at present different models of care to deliver healthcare for the screening and management of comorbidities for PLWH. Fully integrated care of both HIV and comorbidities in a one-stop clinic brings numerous benefits, including optimal utilization of resources, provision of holistic care, and de-stigmatization; but also encounters various challenges, such as placing burden on human and spatial resources in HIV clinics, and the limited availability of co-medications in HIV clinics. In high-income settings, traditional models of care are often physician-centred, thus more innovative models have been explored, involving integrated care in the primary care setting, or consultations by multiple specialists in an integrated clinic, but these require a high magnitude of coordination and have resource implications, limiting feasibility universally. On the other hand, a "differentiated service delivery (DSD)" model is an adaptive model of care that aims to tailor healthcare delivery services according to patients' individual clinical needs and preferences, while taking into consideration resource availability in the local context. This model of care is successful in the delivery of HIV care and management of ART, and is patient-centred, offering patients a mode of care most optimal for their lifestyle and needs without imposing unmanageable burden on the healthcare system. DSD is advocated to be developed for the aging population of PLWH to provide patient-centred healthcare service for management of their comorbidities and other age-related issues, but has not been well studied.

The rising use of telemedicine since the Coronavirus disease 2019 (COVID-19) pandemic in the management of HIV and other chronic diseases would facilitate the incorporation of more patient-centred options in healthcare service delivery according to patients' needs and preferences. Telemedicine interventions improve access to care, control of disease, and quality of life in people with chronic non-communicable diseases. In particular, telemonitoring interventions and synchronous video teleconsultations are found to be beneficial in disease control and enhancing patient-physician interaction.

The currently proposed DSD model of care has the following benefits: (1) patient-centred care with individualized care delivery options according to patients' preference, such as offering teleconsultation as an alternative, options of different drug delivery modes, and personalized management plans according to individual clinical needs; (2) shared care between HIV care providers and internal medicine specialists, with close communication regarding clinical data and treatment plans, while avoiding duplication of resources; (3) draws on the availability of telemedicine tools in public healthcare services in Hong Kong; (4) patient empowerment by educating patients on treatment goals, performing selfmonitoring of disease, and scheduling appointments according to clinical indications; and (5) optimizing care of complex comorbidities by providing specialist care, and screening and management of comorbidities according to evidencebased guidelines.

ELIGIBILITY:
Inclusion Criteria:

* PLWH eligible to participate in this study are PLWH aged 18 years or above
* followed up at the HIV Clinic, and with one or more cardiometabolic comorbidities, including hypertension, diabetes, hyperlipidaemia, metabolic-associated fatty liver disease, cardiovascular diseases, and cerebrovascular diseases. They will be eligible if HIV physicians consider them having sub-optimal control of their comorbidities, suspected of having complications, or would benefit from screening of complications resulting from their comorbidities. These indications are selected as they involve specialist care, including investigations and treatment, which are not available at the HIV Clinic.

Exclusion Criteria:

* Incompetent subjects who cannot give informed written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PLWH eligible to participate in this study are PLWH aged 18 years or above followed up at the HIV Clinic, and with one or more cardiometabolic comorbidities, including hypertension, diabetes, hyperlipidaemia, metabolic-associated fatty liver disease, cardiovascular diseases, and cerebrovascular diseases.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of PLWH | Baseline
  Acceptability of PLWH, as defined by the proportion of PLWH who perform the survey who indicate "willingness to participate" in the DSD programme.
Participation willingness | Baseline
  Similarities and differences between PLWH who are willing and not willing to participate in the DSD programme, by comparing their demographic and clinical data, and the factors assessed in the survey that are associated with perceived benefits and barriers to participation in this programme

SECONDARY OUTCOMES:
Impact on clinical outcomes | At 12 months
  Number of new diagnoses made and changes in ART regimen per 100 patient-year follow-up during participation of the Programme, compared with the same parameters in the 12 months preceding the participation in this Programme.
Unscheduled clinic visits | 12 months preceding the participation in this Programme
  Safety is measured by the number of unscheduled clinic visits at general out-patient clinics, ad hoc HIV clinic telephone enquiry and consultations, Accidents and Emergency Department attendance, and hospital admission per 100 patient-year follow-up during participation of the Programme, compared with the same parameters in the 12 months preceding the participation in this Programme
Satisfaction with the Programme among PLWH | At 12 months
  Satisfaction is defined by the level of satisfaction with the Programme among PLWH. This is measured by a survey to be administered at the end of 12 months follow-up, to determine level of satisfaction with each of the components of the Programme and overall satisfaction.
Changes in systolic and diastolic blood pressure | Through study completion, an average of 1 year
  Changes in systolic and diastolic blood pressure during study.
Changes in body weight | Through study completion, an average of 1 year
  Changes in body weight during the study.
Changes in body mass index | Through study completion, an average of 1 year
  Changes in body mass index during the study
Changes in fasting glucose | Through study completion, an average of 1 year
  Changes in fasting glucose during the study
Changes in HbA1C | Through study completion, an average of 1 year
  Changes in HbA1c during the study
Changes in lipid profiles | Through the study completion, an average of 1 year
  Changes in lipid profiles such as total cholesterol, LDL cholesterol, HDL cholesterol and triglyceride during the study
Changes in creatinine | Through study completion, an average of 1 year
  Changes in creatinine during the study
Changes in alanine transaminase | Through study completion, an average of 1 year
  Changes in alanine transaminase during the study
Self-reported adherence to non-ART medications | Through the study completion, an average of 1 year
  Adherence to prescribed non-ART medications is measured by self-reported adherence to prescribed non-ART medications in the preceding 7 days of the consultations.
Change in health-related quality of life (HrQoL) measured by SF12 | Through study completion, an average of 1 year
  Change in health-related quality of life (HrQoL) measured by SF12 during the study
Change in health-related quality of life (HrQoL) measured by WHOQOLHIV BREF | Through study completion, an average of 1 year
  Change in health-related quality of life (HrQoL) is measured by WHOQOLHIV BREF during the study
Preception by healthcare workers at HIV clinic | This survey will be performed at baseline and after all patients completed all follow-ups.
  Perception of this programme as a whole, and its key components, as agreeable or not. Healthcare workers at the HIV clinic will be asked to complete a survey for assessment of their perception of the programme and intention to refer eligible patients to the Programme. This survey will be performed after the Briefing session at HIV clinic, and after completion of all participant recruitment.
  Factors which healthcare workers anticipate or have encountered that are facilitators and barriers to refer eligible patients to the Programme will be evaluated from the survey.
Feasibilty 1- Rate of recruitment | At 12 months
  Recruitment rate is defined as the proportion of PLWH attending the first consultation at the Comorbidities Clinic among all PLWH who have participated in the Acceptability Survey.
Feasibilty 2- Retention rate of the Programme | At 12 months
  Retention rate of the Programme is defined as the proportion of PLWH completed 12-month follow up among those agreed to join the Programme.
Fidelity 1 | At 12 months
  Fidelity is defined as the extent to which the Programme is conducted as planned in our original protocol, including adherence to the protocol and quality of programme delivery. Adherence to each core component of the Programme is assessed, and is defined as the proportion of PLWH completing all complication screening procedures
Fidelity 2 | At 12 months
  Fidelity is defined as the extent to which the Programme is conducted as planned in our original protocol, including adherence to the protocol and quality of programme delivery. Adherence to each core component of the Programme is assessed, and is defined as the proportion of scheduled teleconsultations attended by PLWH
Fidelity 3 | At 12 months
  Fidelity is defined as the extent to which the Programme is conducted as planned in our original protocol, including adherence to the protocol and quality of programme delivery. Adherence to each core component of the Programme is assessed, and is defined as the proportion of teleconsultations with prior submission of report from eHealth Management module
Fidelity 4 | At 12 months
  Fidelity is defined as the extent to which the Programme is conducted as planned in our original protocol, including adherence to the protocol and quality of programme delivery. Adherence to each core component of the Programme is assessed, and is defined as the proportion of PLWH who have co-medications delivered according to opted mode of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Grace LUI, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No